CLINICAL TRIAL: NCT01435694
Title: The Effects of Robot-assisted Gait Training on Locomotor Function and Motor Unit Firing in Multiple Sclerosis Subjects With Severe Gait Impairments. A Randomized Control Trial
Brief Title: Robot-assisted Gait Training in Multiple Sclerosis Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FISM_grant_2010
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; gait rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted gait training (Experimental): Subjects will wear a harness attached to a system to provide body weight support and they will walk on a treadmill with the help of a robotic-driven gait orthosis. The legs are guided according to a physiological gait pattern. The torque of the knee and hip drives can be adjusted from 100% to 0% for one or both legs. The speed of the treadmill can be adjusted from 0 km/h to approximately 3 km/h and body weight support from 0% to 100%. Training sessions will last for an hour with 30 minutes of real walking time, because subject set-up in the device take approximately 30 minutes.
  Interventions: Behavioral: Lokomat (Hocoma, Switzerland)
- Conventional Therapy (Active Comparator): Training sessions will focus on locomotor function improvements. Subjects will receive 45 minutes of individual conventional physiotherapy for session. During the first 5-10 minutes the subjects will perform lower-limb and core stretching exercises to increase muscles flexibility; then they'll deal with lower-limb muscles strengthening exercises tailored on their baseline characteristics (10 minutes). After that they will be trained on walking abilities (like walking at different speeds, rapid changes directions) for 30 minutes with or without assistive aids.
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Lokomat (Hocoma, Switzerland)
  Other Names: robotic-driven gait orthosis
  Arms: Robot-assisted gait training
Behavioral: Conventional Therapy
  Arms: Conventional Therapy

SUMMARY:
Aims of the study:

This is a randomized-controlled trial to test the effects of robot-assisted gait training on locomotor function and motor unit firing rate in multiple sclerosis subjects with severe gait impairments. The control group will be treat with conventional physical therapy.

Subjects and methods:

60 multiple sclerosis patients will be recruited in two outpatient rehabilitation clinics.

Informed consent will be obtained. Participants will be randomized to Robot-assisted gait training (experimental group) or conventional therapy (control group) through a randomization stratification approach, according to a block randomization of 4.

The experimental group will receive 12 robot-assisted gait training sessions over 6 weeks (2 sessions/week). The control group will receive 12 conventional therapy sessions over 6 weeks (2 sessions/week), that will focus on gait training.

Primary outcome measures will be both neurophysiological measures (motor unit firing rate characteristics) and clinical test for gait speed (10m walking test). Secondary outcome measures will include: clinical tests of walking endurance (six minute walking test), balance (Berg Balance Test) and mobility (Up and Go Test).

Clinical assessment of lower-extremities spasticity (Modified Ashworth Scale), motor fatigue (Fatigue Severity Scale), depression (PHQ-9) and quality of life (SF-36) will be monitored. Subject acceptance and confidence in the treatments will be track with a Visual Analog Scale. Outcome measures will be assessed the week prior to treatment initiation (T0), after 6 sessions (T1), the week after the end of treatment (T2) and at 3 months follow-up (T3) to evaluate treatments retention, by a clinician blinded to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* males and females, community dwelling, age 18 or older
* diagnosis of multiple sclerosis in a stable phase, with relapses > 6 months prior to study enrollment
* moderate to severe gait impairments referred to Expanded Disability Status Scale (EDSS) between 6 and 7

Exclusion Criteria:

* neurologic conditions in addition to multiple sclerosis that may affect motor function
* medical conditions likely to interfere with the ability to safely complete the study
* impaired cognitive functioning: Mini Mental Status Examination < 24
* severe lower-extremities spasticity or contractures that may limit range of motion(Ashworth score >4 for hip, knee or ankle flexors/extensors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
motor unit firing rate characteristics | 12 months
  It will be performed through the analysis of superficial EMG signals during isometric knee extension.

SECONDARY OUTCOMES:
walking endurance | 12 months
  six minute walking test
mobility | 12 months
  Timed Up and Go Test
balance | 12 months
  Berg Balance Test
gait speed | 12 months
  10 meter test
Fatigue | 12 months
  Fatigue Severy Scale
quality of life | 12 months
  SF-36
depression | 12 months
  patient health questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Study Chair — Ferrara University Hospital; Carmelo Chisari, MD, Study Chair — Pisana University Hospital; Nino Basaglia, MD, Principal Investigator — Ferrara University Hospital
Locations (1):
- Physical Medicine and Rehabilitation Department, Ferrara, Ferrara, Italy